CLINICAL TRIAL: NCT01012206
Title: Overweighed Children´s Health - Studies of the Effect of Lifestyle and Food Habits
Acronym: SELFH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Christel Larsson, Professor, Göteborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05-088M
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Overweight; Obesity
Keywords: Children; Overweight; Obesity; Food habits; Dietary assessment; Physical activity
MeSH Terms: conditions — Overweight; Obesity; Feeding Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Children in control group obtained no lifestyle counseling (intervention).
- Intervention group (Active Comparator): Children in the intervention group and their parents were given lifestyle counseling and participated in an intervention program regarding food habits and physical activity.
  Interventions: Behavioral: Intervention regarding food habits and physical activity.

INTERVENTIONS:
Behavioral: Intervention regarding food habits and physical activity. — Children in the intervention group participated in an intervention program regarding food habits and physical activity.
  Arms: Intervention group

SUMMARY:
The aim is to investigate the development of overweight and obesity from infancy to school age, and to evaluate an intervention to prevent further development of overweight and obesity among children.

A follow-up study will be conducted on 267 children and will allow comparison between children that developed overweight with the ones who did not. Subjects will be requited at 10 years of age from a previous project. These children have been studied when they were 6-18 months old and a follow-up was conducted at 4 years of age. Sixteen percent of the children were overweight at 4 years of age and retrospective data of e.g. food intake, blood lipids and anthropometric measurements exists. In the present follow-up data regarding food and physical activity habits, anthropometric measurements and blood samples of e.g. blood lipids, IGF1 will be collected.

An intervention study will be conducted on 80-120 overweight children that will be randomized into one intervention and one control group. An intervention during two years will encourage long term healthy habits regarding diet and physical activity through group meetings and supervision. Information about food habits will be collected through questionnaires, interviews and diaries. Measurement of physical activity and energy expenditure will be made with Sense Wear and double labeled water, and will be used to validate reported food intake. Further, anthropometric measurements and blood samples will be collected.

ELIGIBILITY:
Inclusion Criteria for SELFH intervention study:

* age and gender adjusted body mass index (BMI) > 25
* born in 1995-1998
* living in or nearby the northern city of Umea, Sweden

Exclusion Criteria for SELFH intervention study:

* no chronic disease that could influence metabolic parameters
* no attention deficit disorders
* no access to internet

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2006-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | Two years

SECONDARY OUTCOMES:
Food intake | Two years
Physical activity | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Christel Larsson, PhD, Principal Investigator — Department of Food and Nutrition, Umeå university.
Locations (1):
- Umeå university, Umeå, Sweden

REFERENCES:
- [Result] Waling MU, Larsson CL. Energy intake of Swedish overweight and obese children is underestimated using a diet history interview. J Nutr. 2009 Mar;139(3):522-7. doi: 10.3945/jn.108.101311. Epub 2009 Jan 21. PMID 19158227